CLINICAL TRIAL: NCT04246424
Title: Randomized Experiment of Sleep Technology Study
Brief Title: Randomized Experiment of Sleep Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kelly Glazer Baron, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00117330
Record Dates: First submitted 2019-12-10; First posted 2020-01-29 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fitbit + Coaching (Active Comparator): Fitbit + coaching will receive both the fitbit and coaching interventions.
  Interventions: Behavioral: Fibit + Coaching
- Coaching (Active Comparator): Coaching group will receive weekly remote coaching lessons by phone email or text for 1-6 weeks. They will also receive a weekly email lesson for 1-6 weeks on things such as basics of sleep, enhancing sleep environment and managing stress.
  Interventions: Behavioral: Coaching
- Fitbit (Active Comparator): Fitbit group will receive a Fitbit and are asked to monitor their sleep over the smartphone application for 1-6 weeks.
  Interventions: Behavioral: Fitbit
- Self-management (No Intervention): Self-management participants will be given some information of improving sleep but asked to keep their same schedule. Once their participation concludes, they will be given the opportunity to receive a fitbit and coaching if they so choose.

INTERVENTIONS:
Behavioral: Fibit + Coaching — This intervention is a combination of the coaching and fitbit interventions
  Arms: Fitbit + Coaching
Behavioral: Coaching — Coaching Participants who are assigned coaching group will receive telephone coaching. Coaches follow a guide developed by Kelly Glazer Baron, Jennifer Duffecy, Kathryn Reid, and Lauren Caccamo. The first session is an approximately 30 minute engagement session, with the purpose of "getting to know" the participant to increase likelihood for participation. The end goal is to have participants express Desire, Ability, Reason, Need, Can (DARN-C) to make changes in sleep). The remainder calls (week 2-6) are follow-up calls lasting about 5 minutes. The goal of these calls is to keep participants motivated and address any issues with the Fitbit hard or software.
  Participants will also receive weekly email lessons to their personal email address for 1-6 weeks.
  Arms: Coaching
Behavioral: Fitbit — Fitbit Participants in the fitbit group will receive a Fitbit Charge 3 black, and asked to wear it for 1-6 weeks. Participants will monitor their sleep through the sleep section in the Fitbit app on the smartphone. Participants will be provided login information so that researchers can access this data and asked to keep Bluetooth on. After week 6, participants can choose to continue to wear the device for the duration of the study (12 weeks). Though wear at weeks 7-12 is not required, researchers will still use any data that was collected from the fitbit during that time. At the completion of their participation, researchers retain the login information and the device is switched to a personal login of the participants choice.
  Arms: Fitbit

SUMMARY:
Short sleep duration is highly prevalent and linked to negative mental and physical health consequences, including increased cardiovascular disease risk [1]. According to data from the National Health Interview Survey, 70.1 million U.S. adults (29.2%) sleep <6 hours per 24 hour period [2]. These statistics are a stark contrast to recommendations made by a recent consensus panel of sleep experts that concluded "at least 7 hours" is the amount of sleep needed for health and performance among adults [3]. Therefore, a high number of U.S. adults could benefit from extending sleep duration. Several small experiments have demonstrated the benefits of short-term sleep extension [4-8]. However, these studies are limited by extending sleep as a temporary experimental manipulation rather than a longer-term behavioral intervention. To deliver sleep extension interventions, wearable sleep trackers may be useful, particularly given the rapid uptake among consumers (+500% in 3 years) [9]. We have developed a novel technology-assisted behavioral sleep extension intervention that employs four elements -- a wearable sleep tracker, didactic content, an interactive smartphone feature and brief telephone counseling. User testing supports feasibility of extending sleep, but little is known about the effects of differing types of technology interventions on sleep. Therefore, the goal of this study is to examine the differences between technology sleep extension interventions and sleep duration.

DETAILED DESCRIPTION:
Study Design - Intervention

* Web or phone prescreening: Participants will first complete a brief online screening to determine initial eligibility criteria (self-report of medical and psychiatric conditions, sleep disorders). Individuals who are potentially eligible will be sent an Actiwatch via FedEx, along with training instructions. Participants will wear the Actiwatch for a 7-day prescreening assessment. Research staff will receive verbal consent for this screening procedure and will go over instructions over the phone to ensure participants understand how to use this device.
* Study Visits: Visit 1- Screening assessment: Participants will attend a one hour laboratory visit that will include consent procedures, standardized measurements of height, weight, waist and hip circumference, and blood pressure. Participants will complete baseline study questionnaires.
* Enrollment: During visit 1, staff will review eligibility. Participants will be informed at the end of visit one of their eligibility. If the participant is eligible, they will receive a verbal and written instructions and informing them of their study group assignment. If they are not eligible, a payment will be sent via check.
* Randomization: Participants will be randomized to 4 study groups using sealed envelopes with assignments determined via a random number generator.
* Study Conditions: Participants will be randomly assigned to 1 of 4 study groups.
* Study group 1: Participants will receive the telephone coaching and wear the Fitbit device week 1 through week 6.
* Study group 2: Participants will receive the telephone coaching only.
* Study group 3: Participants will wear the Fitbit device week 1 through week 6 study but will not receive telephone coaching.
* Study group 4: Control group. Participants will not receive telephone coaching nor will they wear the Fitbit device. They will be instructed to keep their sleep schedule consistent.

Arms and Interventions -

* The intervention will be delivered via smartphone and adherence will be facilitated by telephone coaching. Participants will receive weekly "lessons", which are content that is emailed each week as part of the program. In study groups 1 and 3, participants will wear a Fitbit sleep tracking monitor for the duration of the intervention. Coaches will be able to log in and see participants' data to help encourage them to meet their sleep goals.
* Weekly lesson content will be delivered via email (e.g. mail chimp).
* Telephone coaching: Participants in study groups 1 and 2 will be assigned to a sleep coach who will monitor their progress during the study and provide weekly telephone coaching sessions related to their sleep-related goals. The coaches will establish legitimacy by their knowledge of sleep and basic counseling principles. They will establish goals with the participants based on the participants' values and beliefs, including the particular sleep related goals and also usage goals, (e.g., number of log-ins completed per week). Performance monitoring will be completed through an online dashboard visible to the coaches (Fitbit web log in). The first coaching session is a 20 min engagement session, which includes introductions, rational for the program, clarifying roles of the coach and the participants' goals for the program. Coaches (directed by Dr. Baron) will provide feedback to the participant based on Fitbit and sleep diary data. For weeks 2-6, the coach and participant will also have weekly brief (5-10 min) follow-up support calls to troubleshoot any problems with the application or Fitbit, review progress, problem solve barriers to progress, and set goals for the following week. In-between sessions, the coaches will be available, mostly over email, to troubleshoot any problems with the content or Fitbit. Frequency of text, phone, and email communication will be recorded.
* Control group: Participants assigned to the no-treatment wait list control condition will be told they were assigned to the wait list group, and therefore eligible to receive the intervention components at the end of the study. At the end of the final session, they will receive a Fitbit wearable fitness tracker and emails with the 6 didactic lessons.

ELIGIBILITY:
Inclusion Criteria:

1. BMI >25 kg/m2
2. Short sleep duration (<6.5 hrs of sleep per night, on average)

Exclusion Criteria:

1. High risk or presence of restless legs syndrome or insomnia as assessed by the screening questionnaires,
2. History of cognitive or neurological disorders;
3. Presence of any major psychiatric disorder, current alcohol or substance abuse;
4. Unstable or serious medical illness;
5. Shift work or travel over 2 time zones in the past 2 months,
6. Inability to read and write English,
7. Pregnancy or desire to become pregnant during the study period,
8. Significant environmental factors disturbing sleep (e.g. awakenings >4 per week due to caregiving responsibilities),
9. >8 hours in bed on average,
10. engaged in special diet for weight loss (e.g., diet post weight loss surgery),
11. use of hypnotics within the past three months.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Sleep Duration (Assess changes in sleep quality) | time points at visit 1 (week 1), visit 2 (week 6) and visit 3 (week 12)
  Assess changes in sleep quality:Using the Philips Respironics Actiwatch (scoring completed using Philips Actiware 6), sleep duration and sleep quality will be assessed. Measures include bed/wake time, total time in bed, total sleep time, onset latency, sleep efficiency, number of awakenings and minutes awake during the night, or Wake After Sleep Onset (WASO). White, red, green and blue light will be measured using the device but only white light will be used in the assessment.
Sleep Duration | time points at visit 1 (week 1), visit 2 (week 6) and visit 3 (week 12)
  Assesses changes in daytime sleepiness: Using questionnaires Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment (2008-2012 PROMIS Health Organization and PROMIS Cooperative Group)
Sleep Duration | time points at visit 1 (week 1), visit 2 (week 6) and visit 3 (week 12)
  Assesses changes in daytime sleepiness: Munich Chronotype Questionnaire (Chronotype(en) 2008 Till Roenneberg, & Martha Merrow, LMU Munich) , daytime sleepiness and changes over the three time points will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Family and Preventive Medicine, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided